CLINICAL TRIAL: NCT04642092
Title: Treatment for Emotional Disorders in Primary Care Units With Evidence-Based Psychological Techniques and mHealth: A Randomized Controlled Trial
Brief Title: Evidence-Based Psychological Treatment for Emotional Disorders Attended in Dominican Primary Care Units (PsicAP)
Acronym: PsicAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica Madre y Maestra (Other)
Collaborators: Ministerio de Educación Superior, Ciencia y Tecnología, Dominican Republic (Unknown)
Responsible Party: Principal Investigator, Zoilo Emilio García Batista, PhD in Cognition, Emotion and Health; Director of the Vice-Rectory of Research and Innovation in PUCMM, Pontificia Universidad Catolica Madre y Maestra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-2019-2A1-96
Record Dates: First submitted 2020-10-12; First posted 2020-11-24 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Anxiety Disorders; Depression; Somatic Disorders; Emotional Disorder
Keywords: Cognitive Behavioral Therapy; Primary Care; Emotional Disorders
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and therapists will know if they are from the control or the experimental group. This study will be blinded only for the evaluators (the ones who will apply the psychological tests). Psychologists with the the role of evaluators will not give any therapy to the participants, and will not know from which group the patients are, neither who gave them the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PsicAP protocol (Experimental): The treatment of the experimental group will be according to the PsicAP protocol: seven sessions of a psychological treatment based on transdiagnostic approaches, collaborative interventions, group-sessions, and evidence-based psychological techniques derived from cognitive behavioral therapy.
  Interventions: Behavioral: PsicAP protocol
- Conventional treatment (Active Comparator): The control group will have seven sessions based on the typical psychological services that currently are offered in the Dominican Primary Care Units.
  Interventions: Behavioral: Conventional treatment

INTERVENTIONS:
Behavioral: PsicAP protocol — The intervention will include: psychoeducation, relaxation and breathing techniques, thought management, tips to improve quality of life and relapse prevention. All of these activities will be based on scientific evidence and many of these aspects will be supported by mobile devices.
  Other Names: Evidence-Based Psychological Techniques and mHealth
  Arms: PsicAP protocol
Behavioral: Conventional treatment — Typical treatment that is currently given to patients with emotional disorders in Dominican primary care units.
  Arms: Conventional treatment

SUMMARY:
Emotional disorders affect millions of people all over the world. Thousands of Dominicans suffer from depression, anxiety, and other emotional disorders that have negative impact on their lives. Nevertheless, many of them do not receive a proper treatment. The purpose of this study is to describe a pilot project, in which a protocol of evidence-based psychological treatment for emotional disorders, supported by mHealth (mobile health), will be applied on Dominicans who attend Primary Care services. It will be a collaborative program, divided into three phases, and based on cognitive behavioral therapy. The hypothesis of this research is that this protocol is an effective strategy to treat emotional disorders.

DETAILED DESCRIPTION:
Emotional disorders, such as anxiety, depression and somatic disorders, represent a serious public health issue. Many people who suffer from them do not have access to an adequate psychological treatment. Some of the reasons why this situation happens are: the high cost that tends to represent a proper psychological treatment, and, in countries like Dominican Republic, the lack of a protocol that guides health professionals of Primary Care Units on the diagnosis and treatment of these emotional disorders. The purpose of this study is to describe a pilot project, in which a treatment protocol for emotional disorders will be applied by trained mental health professionals in Dominican Primary Care Units. It will be a randomized controlled trial with 300 patients. To prove the effectiveness of this protocol, the phases of this study will be: 1) psychological assessment of the study sample; 2) seven sessions of conventional treatment offered to a control group, and seven sessions of the evidence-based psychological techniques, suggested by this new protocol, given to an experimental group; 3) psychological reassessment of the study sample. This protocol suggests transdiagnostic approaches and collaborative interventions, that include group-sessions and evidence-based psychological techniques derived from cognitive behavioral therapy. Also, the protocol will be supported by mHealth tools. Some of the points included in the protocol are: psychoeducation on emotional disorders symptoms, relaxation and breathing techniques, thought management, improvement of quality of life and relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 79 years old.
* Adults with mild or moderate levels of anxiety, depression or somatic disorders.
* Dominicans.
* People who are not receiving any psychological treatment.
* People who know how to read and write.

Exclusion Criteria:

* A diagnostic of severe mental/emotional disorder.
* Recent suicide attempt.
* Severe disability.
* People who do not meet sufficient criteria to be diagnosed with mental or emotional disorders.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in the score of Patient Health Questionnaire-2 | An average of 16 months (from baseline to psychological treatment completion).
  On Patient Health Questionnaire-2 (PHQ-2), patients are asked how often, in the last two weeks, they have been bothered by depressed mood and anhedonia. Each response option is scored from 0 to 3. Therefore, total scores of the scale range from 0 to 6. A score of 3 or greater means high possibility of major depressive disorder.
Change in the score of Patient Health Questionnaire-4 | An average of 16 months (from baseline to psychological treatment completion).
  On Patient Health Questionnaire-4 (PHQ-4), subjects are asked how often, in the last two weeks, they have been bothered by core symptoms/signs of depression and anxiety. This test has two subscales: one of them has two items that evaluate depression; the other one, two items that assess anxiety. Each response option is scored from 0 to 3, so total scores for each subscale range from 0 to 6. A score of 3 or greater on the depression subscale represents a high probability of this disease; a score of 3 or greater on the anxiety subscale means that the prevalence of an anxiety disorder is likely.
Change in the score of Patient Health Questionnaire-9 | An average of 16 months (from baseline to psychological treatment completion).
  On Patient Health Questionnaire-9 (PHQ-9), through 9 items, subjects are asked how often, in the last two weeks, they have been bothered by core symptoms of depression. Each response option is scored from 0 to 3, so total scores range from 0 to 27. PHQ-9 scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively.
Change in the score of Patient Health Questionnaire-15 | An average of 16 months (from baseline to psychological treatment completion).
  On Patient Health Questionnaire-15 (PHQ-15), through 15 items, subjects are asked how often, in the last 4 weeks, they have been bothered by somatic symptoms. Each response option is scored from 0 to 2. Therefore, total scores range from 0 to 30. PHQ-15 scores of 5, 10, 15, represent cutpoints for low, medium, and high somatic symptom severity, respectively.
Change in the score of Patient Health Questionnaire-PD | An average of 16 months (from baseline to psychological treatment completion).
  The Patient Health Questionnaire-Panic Disorder (PHQ-PD) is actually a section of PHQ, which comprises 15 items (questions 3a-d and 4a-d-k are the ones that evaluate PD). There are two answer categories: "no" (0 points) and "yes" (1 point.). Therefore, total scores range from 0 to 15. In Spanish population, the best cutoff score for screening panic disorder in patients is 5.
Change in the score of Generalized Anxiety Disorder Test-2 | An average of 16 months (from baseline to psychological treatment completion).
  On Generalized Anxiety Disorder Test (GAD-2), through two items, subjects are asked how often, in the last two weeks, they have been bothered by core symptoms of anxiety. Each response option of the scale is scored from 0 to 3, so total scores range from 0 to 6. GAD-2 score of 3 represent the best cutoff point for screening generalized anxiety disorder.
Change in the score of Generalized Anxiety Disorder Test-7 | An average of 16 months (from baseline to psychological treatment completion).
  On Generalized Anxiety Disorder Test-7 (GAD-7), through seven items, subjects are asked how often, in the last two weeks, they have been bothered by core symptoms of generalized anxiety disorder. Each response option of the scale is scored from 0 to 3, so total scores range from 0 to 21. Scores of ≥5, ≥10, and ≥15 represent mild, moderate, and severe anxiety symptom levels, respectively.
Change in the score of Sheehan Disability Inventory | An average of 16 months (from baseline to psychological treatment completion).
  The Sheehan Disability Inventory (SDS) is a 5-item self-report tool. In the first three items, patients rate their functional impairment in work/school, social life, and family life, by a 10-point visual analog scale in each case. Scores of ≥5 on any of the three scales are associated with significant functional impairment. The last two items evaluate the amount of days lost or unproductive due to the functional impairment.
Change in the score of the Brooding subscale from Ruminative Responses Scale (RRS) | An average of 16 months (from baseline to psychological treatment completion).
  The Ruminative Responses Scale (RRS) has 22 items. Patients must indicate what they generally do when they feel down, sad, or depressed, using a 4-point Likert-type scale representing frequency (1=never; 4=always). The brooding subscale is composed by 5 of the 22 items of the whole scale. Therefore, total scores of this subscale range from 5 to 20. Higher scores on this subscale indicate significant levels of brooding.
Change in the score of the Penn State Worry Questionnaire (PSWQ) | An average of 16 months (from baseline to psychological treatment completion).
  The Penn State Worry Questionnaire (PSWQ) is a 16-item questionnaire. Items are rated using a 5-point Likert-scale (from 1="not at all typical of me" to 5="very typical of me"). Therefore, total scores range from 16 to 80. Scores of ≥16, ≥40, and ≥60 represent low, moderate, and high worry levels, respectively.
Change in the score of Inventory of Cognitive Activity in Anxiety Disorders | An average of 16 months (from baseline to psychological treatment completion).
  Inventory of Cognitive Activity in Anxiety Disorders (IACTA; Inventario de Actividad Cognitiva en los Trastornos de Ansiedad) is an instrument that evaluates certain cognitive activity in patients with different types of anxiety disorders. It has three subscales: panic attack (14 items), agoraphobia (14 items), and social phobia (20 items). Subjects are asked to indicate how often they pay attention to certain cognitive distortions about symptoms related to those disorders, ranging from 0 (almost never) to 4 (almost always). Higher the scores, higher the probability of suffering from a type of anxiety disorder. A cutoff point of 48 on panic attack and agoraphobia subscales was related to the prevalence of panic disorder; a cutoff point of social phobia subscale was related to suffering from social phobia disorder.
Change in the score of Questionnaire of Cognitive Distorsions in Emotional Disorders | An average of 16 months (from baseline to psychological treatment completion).
  Questionnaire of Cognitive Distorsions in Emotional Disorders (CDTE; Cuestionario de Distorsiones Cognitivas en los Trastornos Emocionales) is an instrument that evaluates the frequency with which certain cognitive distortions appear. It has 52 items. Each response option of the scale is scored from 0 (almost never) to 4 (almost always). Therefore, total scores range from 0 to 208. Higher scores indicate greater levels of cognitive distortions.
Change in the score of Emotion Regulation Questionnaire (ERQ) | An average of 16 months (from baseline to psychological treatment completion).
  Emotion Regulation Questionnaire (ERQ) is a 10-item scale that measures patients' tendency to regulate their emotions in two ways: cognitive reappraisal and expressive suppression. Each response option is scored by a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). Therefore, total scores range from 10 to 70. The higher the score, the greater the use of emotion regulation strategies.
Change in the score of Metacognitions Questionnaire (MCQ-30) | An average of 16 months (from baseline to psychological treatment completion).
  Metacognitions Questionnaire (MCQ-30) measures individual differences in meta-cognitive beliefs, judgments and monitoring tendencies. It comprises a total of 30 items. Responses to each item are based on a 4-point Likert scale (from 1 = "do not agree" to 4 = "strongly agree"). MCQ-30 scores range from 30 to 120 points. Higher scores indicate greater pathological meta-cognitive activity.
Change in the score of World Health Organization Quality of Life - BREF (WHOQOL-BREF) | An average of 16 months (from baseline to psychological treatment completion).
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire that evaluates four domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. In addition, there are two items that measure overall QOL and general health. The whole scale is formed by 26 items. Subjects have to answer according to how they have been feeling in the last two weeks. Responses to each item are based on a 5-point Likert scale (from 1 = "not at all" to 5 = "completely"). The raw score ranges of each domain are: 7-35 for physical health, 6-30 for psychological health, 3-15 for social relationships, and 8-40 for environment. Higher scores denote higher quality of life.
Change in the score of EuroQol-5 D (EQ-5D) | An average of 16 months (from baseline to psychological treatment completion).
  EuroQoL is an instrument that measure the quality of life related to health. It has two main parts. The first part is a descriptive system in which subjects indicate how they feel, during the current day of the assessment, in the following areas of their lives: movement ability, personal care, daily activities, pain and anxiety/depression. Responses to each item are based on three options: 1 (no problems), 2 (some/moderate problems), 3 (many problems). Higher scores on these items denote worse quality of life. The second part is a visual analog scale in which subjects must indicate how they evaluate their health condition during the current day of the evaluation (from 0=the worst health condition, to 100=the best health condition).

CONTACTS AND LOCATIONS:
Overall Officials: Zoilo E García Batista, PhD, Principal Investigator — Pontificia Universidad Catolica Madre y Maestra; Kiero Guerra Peña, PhD, Study Chair — Pontificia Universidad Catolica Madre y Maestra; Antonio Cano-Vindel, PhD, Study Chair — Universidad Complutense de Madrid; Ricardo Araya, PhD, Study Chair — King's College London
Locations (4):
- Dominican Republic (4):
  - Centro de Atención Primaria Dr. Sergio Bisonó (Barrio Lindo), Santiago de los Caballeros, Santiago Province
  - Centro de Atención Primaria El Guano, Santiago de los Caballeros, Santiago Province
  - Centro de Atención Primaria Mamachen, Santiago de los Caballeros, Santiago Province
  - Centro Diagnóstico Gurabo, Santiago de los Caballeros, Santiago Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cano Vindel A. Bases teóricas y apoyo empírico de la intervención psicológica sobre los desórdenes emocionales en Atención Primaria. Una actualización. Ansiedad y estrés. 2011; 17(2-3): 157-184.
- [Derived] Garcia-Batista ZE, Cantisano-Guzman LM, Guerra-Pena K, Alvarez A, Moretti L, Cano-Vindel A, Munoz-Navarro R, Medrano LA, Baltra RA. PsicAP transdiagnostic protocol of group cognitive-behavioral training for emotional disorders in Dominican Republic: a randomized controlled trial protocol. BMC Psychiatry. 2023 May 24;23(1):363. doi: 10.1186/s12888-023-04771-3. PMID 37226144